CLINICAL TRIAL: NCT01640717
Title: A Retrospective, Observational, Noninterventional Data Collection Study for Patients With Molybdenum Cofactor Deficiency Who Have Been Previously Treated With Cyclic Pyranopterin Monophosphate (cPMP)
Status: Completed | Type: Observational
Sponsor: Origin Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-MCD-501; ALX-MCD-501 (Registry Identifier: ALX-MCD-501)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Molybdenum Cofactor Deficiency
MeSH Terms: conditions — Molybdenum cofactor deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to assess safety and efficacy data of Escherichia coli-derived cPMP in patients with molybdenum cofactor deficiency (MoCD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any age.
2. Patient with MoCD type A, suspected type A, or type B.
3. Patient previously received cPMP only by intravenous route of administration.
4. Parent(s) or legal guardian(s), depending on local regulations, has voluntarily provided written informed consent for the Investigator, Investigator's designee, or Sponsor designee to review, collect, transmit, and analyze data extracted from the medical record. In the case of a deceased patient for whom the parents or legal guardians could not be located, the appropriate ethical review committee may assign another person as legal representative to provide consent, where applicable per local and country regulations.

Exclusion Criteria:

* Patient's parent(s) or legal guardian(s) are unable to understand the nature and scope of the study.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received only intravenous cPMP under named-patient use will be eligible
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy | For up to 60 months from the initial date of treatment with cPMP
  This is a noninterventional, observational, retrospective study to collect data on pediatric patients with MoCD who have received E. coli derived cPMP by intravenous only administration. The study will neither provide treatment with cPMP nor alter any ongoing treatment schedules; rather, its objective is to retrospectively collect data on MoCD history and previous treatment with intravenous E. coli derived cPMP, which is documented in the medical records of patients who have received treatment according to a named patient treatment plan.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Neonatologist, Department of Paediatrics, Mercy Hospital for Women, Heidelberg
  - Monash Medical Centre, Melbourne
  - Western Sydney Genetics Program & Sydney Medical School, Westmead
- Germany (3):
  - University Hospital of Cologne, Cologne
  - Frankfurt Children's Hospital, Frankfurt
  - Akademisches Lehrkrankenhaus der Johannes Gutenberg, Koblenz
- Beatrix Children's Hospital, Groningen, Netherlands
- TC Saglik Bakanligi Gaziantep Cocuk Hastaliklari Hastanesi, Gaziantep, Turkey (Türkiye)
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Royal Hospital for Sick Children, Glasgow
  - Manchester Academic Health Science Centre, Manchester